Protocol At-A-Glance Version 2018.10.18.

Project Title: Hearing Impairment, Strategies and Outcomes in VA Emergency Departments

**Principal Investigator:** Joshua Chodosh, MD, MSHS **Site:** 630 – New York Harbor Healthcare System

## **Study Goals:**

- 1) Establish the feasibility of screening for hearing loss in the ED
- 2) Determine the acceptability of the screening procedure (among ED population)
- 3) Derive a preliminary estimate of effect size of primary outcomes
- 4) Identify the evidence that decision makers in VAMCs, ED and Audiology Services need to commit to this approach

## **Study Outline:**

- -18 month funding period, to include: four month start-up, 12 months of intervention, and two months of analysis, disseminations, and plans for next steps to advance hearing healthcare in VA health system
- -Minimum goal of 68 and maximum is 150 (across both Manhattan and Brooklyn)
- -Patients will be randomized to receiving a HAD or control
- -Data collections from VA CPS, RA observations, 10-minute RA survey, and brief qualitative follow-up interviews with patients, nurses, physicians. Follow-up calls three-days and 30-day ED visits will occur.
- -Brief semi-structured interviews with 10 veterans willing to speak more extensively after discharge from ED
- -Brief semi-structured interviews with 10 nurses and physicians (providers) will access their experiences with the hearing-impaired patients

## Milestones/Developmental Progress Goals (DPGs):

We will track and report on these Milestones regardless of your decision about the feasibility of continued support beyond the 18-month period.

- Hiring and training of research staff
- Successful recruitment of at least 68 subjects who consent to hearing screening in the Emergency Department
- Completion of the HHIE for 85% of consented patients
- Delivery and fitting of the PockeTalker<sup>™</sup> for 85% of patients who score > 10 on the HHIE
- Completion of the HAD use survey for 70% of patients who are given PockeTalkers<sup>TM</sup>
- Completion of the 6-item measure of quality of hearing, understanding, and communication for 70%
- Completion of the CTM-3 for these same 70%
- Successful pilot test of the Patient Understanding of Discharge Instructions (PUDI) for 10 subjects
- Completed semi-structured interviews these 10 subjects and research staff to assess feasibility and refine processes
- Completion of three virtual advisory council meetings with 70% attendance
- Preparation of a summary report of these virtual meetings addressing key issues of feasibility/implementation
- Demonstration of feasibility for all aspects of screening process and delivery, fitting, and teaching PockeTalker<sup>TM</sup> use through observed time/effort, proportion of completed assessments, and patient/provider feedback.

Protocol At-A-Glance Version 2018.10.18.

| Table 5: Project activities and timeline | FY 2018 | | FY 2019 | | | |
|---|---|---|---|---|---|---|
| Tasks: | Q3 | Q4 | Q1 | Q2 | Q3 | Q4 |
| Hiring and training | | | | | | |
| Subject materials preparation | | | | | | |
| Obtain IRB approval | | | | | | |
| Build survey tool | | | | | | |
| Subject recruitment / consent | | | | | | |
| Intervention / usual care study period | | | | | | |
| Subject post-ED visit survey/interview | | | | | | |
| Subject (physician) interviews | | | | | | |
| Medical record data extraction <sup>1</sup> | | | | | | |
| Conduct qualitative analyses | | | | | | |
| Conduct data analyses | | | | | | |
| Write final report | | | | | | |
| Conduct advisory / stakeholder meetings | | | | | | |
| Presentations for dissemination | | | | | | |
| Q1 = Quarter 1, etc | | | | | | |

<sup>&</sup>lt;sup>1</sup>Adminstrative data of all consented subjects on visit and diagnostic variables